CLINICAL TRIAL: NCT03607006
Title: 3D Ridge Augmentation in the Anterior Maxillary Region Using Patient Specific Polyether Ether Ketone (PEEK) Sheets vs. Autogenous Bone Shell Technique. A Randomized Clinical Trial: Comparative Study
Brief Title: Ridge Augmentation Using Patient Specific PEEK Sheets vs. Autogenous Bone Shell Technique.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ola Alaa El-Din Abd El-Monem Mohamed (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Ola Alaa El-Din Abd El-Monem Mohamed, Principle Investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-07-16
Record Dates: First submitted 2018-07-23; First posted 2018-07-31 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Ridge Deficiency
Keywords: Anterior maxillary region; Patient specific; Autogenous bone shell; PEEK; Ridge augmentation

STUDY DESIGN:
Intervention Model Description: * A randomized clinical trial.
  * Parallel group study.
  * A trial will be carried out in hospital of Oral and Maxillofacial surgery department - Faculty of Oral and Dental Medicine - Cairo University .
  * Equal randomization : participants with equal probabilities for intervention.
  * Positive controlled : Both groups receiving treatment.
Masking Description: None because the two interventions requires different preoperative preparations , both the participants and the investigator can't be blinded .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient specific PEEK sheets (Experimental): Patient specific PEEK sheets will be fixed with titanium screws and act as containment system for the mixed autogenous/xenogenic bone graft that will fill the gap between the sheets and the ridge .
  Interventions: Procedure: Patient specific PEEK sheets
- Autogenous bone shell technique (Active Comparator): Bone shells will be fixed with titanium screws to the ridge and mixed autogenous/xenogenic bone graft will fill the gap between the shells and the ridge .
  Interventions: Procedure: Autogenous bone shell

INTERVENTIONS:
Procedure: Patient specific PEEK sheets — Computer aided sheet design
  Arms: Patient specific PEEK sheets
Procedure: Autogenous bone shell — autogenous retromolar/chin bone graft
  Arms: Autogenous bone shell technique

SUMMARY:
Comparative study to assess the ability of the patient specific PEEK sheets in ridge augmentation with using mixed Autogenous/Xenogenic bone graft vs the Bone Shell Technique regarding the time, accuracy and donor site morbidity .

DETAILED DESCRIPTION:
A- Intervention Group (Patient specific PEEK sheets)

* Preoperative Computed tomography will be done to the patients.
* Using special software, 3D models will be obtained and used to design the custom made PEEK sheets. The final STL (Standard Tessellation Language) files will be sent to the lab to be milled/printed.
* Autogenous bone graft will be taken from Chin/Retromolar graft and will be mixed with xenogenic bone graft in 1:1 ratio.
* After bone exposure, the ridge will be decorticated and the prefabricated PEEK sheets will be fixed with titanium screws and the space between the sheets and the ridge will be filled with the prepared bone graft.
* Wounds closure will be done.
* CT scan will be done postoperative.
* After 6 months another CT scan will be done for evaluation and comparison. Then the titanium screws will be removed and implants will be placed.

B- Control Group (Autogenous bone shell technique)

* Preoperative Computed tomography will be done to the patients
* Bone graft will be harvested from the chin/retromolar region and a cortico- cancellous bone block will be obtained then divided into two pieces used as the shells.
* The bone shells will be trimmed and adjusted to the recipient site and the remaining bone will be milled and mixed with Xenogenic bone graft with ratio 1:1
* The bone shells will be anchored in the host bone with titanium screws and the space between the shells and the alveolar bone will be filled by the bone graft mix.
* Wounds closure will be done.
* CT scan will be done.
* After 6 months another CT scan will be done for evaluation and comparison. Then the patient will go for micro screws removal along with implant placement.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with deficient alveolar bone in the anterior maxilla.
* Patient seeking fixed prosthesis at the anterior maxillary region.
* Highly motivated patients.
* Good oral hygiene.
* Patients willing for the surgical procedure and follow-up, with an informed consent.
* Bounded anterior maxilla cases.

Exclusion Criteria:

* Medically compromised patients.
* Uncooperative patients.
* Poor oral hygiene.
* Periodontal diseases.
* No history of any grafting procedure at the designated edentulous ridge.Criteria
* Patients with any diseases that compromise bone or soft tissue healing.
* Patients with no local pathosis that interfere with the bone healing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | 8 months
  Questionnaire will be used to evaluate the satisfaction , measuring unit Binary (YES/NO)

SECONDARY OUTCOMES:
Bone gain | 4-6 months post-operative
  Bone gain will be evaluated using the Computed tomography , measuring unit (mm)
Bone quality | 4-6 months post-operative
  Histological analysis of bone core biopsy , measuring unit Osteon number
Soft tissue reaction | 4-6 months postoperative
  Clinical evaluation by caliber to measure thickness of keratinized mucosa ,measuring unit (mm)
Intraoperative time | Intraoperative
  Using stop watch to measure the operative time

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Brakart, PhD, Study Director — Cairo University; Mohamed M Shaker, PhD, Study Director — Cairo University
Locations (1):
- Faculty of Oral and Dental Medicine - Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mounir M, Morsy OAE, Amer H, Mounir S, Gibaly A. Assessment of bone quality using buccal and palatal autogenous cortical shells harvested from two different mandibular donor sites for maxillary alveolar ridge augmentation: a histomorphometric randomized clinical trial. Oral Maxillofac Surg. 2021 Jun;25(2):263-269. doi: 10.1007/s10006-020-00924-w. Epub 2020 Nov 24. PMID 33231752